CLINICAL TRIAL: NCT05995366
Title: Mass Balance Study of [14C] ABBV-903 in Healthy Male Subjects Following Single Oral Dose Administration
Brief Title: A Study to Assess the Mass Balance of [14C] ABBV-903 in Healthy Male Participants Following Single Oral Dose Administration
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: M24-223
Record Dates: First submitted 2023-08-10; First posted 2023-08-16 (Actual); Last update posted 2023-10-26 (Actual); Status verified 2023-10

CONDITIONS: Healthy Volunteer
Keywords: Healthy Volunteer; ABBV-903

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- ABBV-903 (Experimental): Participants will receive ABBV-903 on Day 1.
  Interventions: Drug: ABBV-903

INTERVENTIONS:
Drug: ABBV-903 — Solution; Oral

SUMMARY:
The purpose of this study is to evaluate the mass balance and safety of [14C] ABBV-903 in healthy male volunteers following a single oral dose administration.

ELIGIBILITY:
Inclusion Criteria:

* Body Mass Index (BMI) is >= 18.0 to <= 32.0 kg/m2 after rounding to the tenths decimal at Screening and upon initial confinement.
* A condition of general good health, based upon the results of a medical history, physical examination, vital signs, laboratory profile and a 12-lead electrocardiogram (ECG).

Exclusion Criteria:

* History: of epilepsy, any clinically significant cardiac, respiratory (except mild asthma as a child), endocrine, metabolic, renal, hepatic, gastrointestinal, Gilbert's Syndrome, hematologic or psychiatric disease or disorder, or any uncontrolled medical illness
* History of any clinically significant illness/infection/major febrile illness, hospitalization, or any surgical procedure within 30 days prior to study drug administration.
* Consider fathering a child or donating sperm during the study and for 94 days after study drug administration.
* Has had significant exposure to radiation for professional or medical reasons (e.g., serial x-rays or computed tomography scans, barium meal, current employment in a job requiring radiation exposure monitoring), except dental x-rays, within 12 months prior to study drug administration.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 7 (Actual)
Dates: Start 2023-08-18 (Actual); Primary Completion 2023-10-13 (Actual); Study Completion 2023-10-13 (Actual)

PRIMARY OUTCOMES:
Maximum observed concentration (Cmax) of ABBV-903 | Up to Day 16
  Cmax of ABBV-903 will be assessed.
Time to Cmax (peak time, Tmax) of ABBV-903 | Up to Day 16
  Tmax of ABBV-903 will be assessed.
Terminal Phase Elimination Half-life (t1/2) of ABBV-903 | Up to Day 16
  Terminal phase elimination half-life (t1/2) will be assessed.
Area Under the Plasma Concentration-time Curve (AUC) from Time 0 to the Time of the Last Measurable Concentration (AUC0-t) of ABBV-903 | Up to Day 16
  AUC0-t of ABBV-903 will be assessed.
AUC from Time 0 to Infinite Time (AUC0-t) of ABBV-903 | Up to Day 16
  AUC0-inf of ABBV-903 will be assessed.
Number of Participants with Adverse Events (AEs) | Baseline to Day 46
  An adverse event (AE) is defined as any untoward medical occurrence in a patient or clinical investigation participant administered a pharmaceutical product which does not necessarily have a causal relationship with this treatment.

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (1):
- Fortrea Clinical Research Unit Inc. /ID# 253962, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — https://www.abbvieclinicaltrials.com/study/?id=M24-223